CLINICAL TRIAL: NCT02905019
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Safety and Protective Efficacy of Adjuvanted R21 at Two Different Doses and the Combination Malaria Vaccine Candidate Regimen of Adjuvanted R21 + ChAd63 and MVA Encoding ME-TRAP.
Brief Title: A Safety and Efficacy Study of R21 +/- ChAd63/MVA ME-TRAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC065
Record Dates: First submitted 2016-07-28; First posted 2016-09-19 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2017-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Matrix-M

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Standard Dose x3 (Group 1) (Active Comparator): R21 with Matrix-M1. Three vaccinations with 10 µg R21/ 50 µg Matrix-M1 on days 0, 28 and 56.
  Interventions: Biological: R21 with Matrix-M1
- High Dose (Group 2) (Active Comparator): R21 with Matrix-M1. Two vaccinations with 50µg R21/50µg Matrix-M1 on days 0 and 28 and one vaccination with 10 µg R21/ 50 µg Matrix M1 on day 56.
  Interventions: Biological: R21 with Matrix-M1
- Combination (Group 3) (Active Comparator): R21 with Matrix-M1, ChAd63 ME-TRAP and MVA ME-TRAP. Three vaccinations with 10 µg R21/ 50 µg Matrix-M1 on days 0 , 28 and 56. Plus one vaccination with ChAd63 ME-TRAP on day 7 and one vaccination with MVA ME-TRAP on day 63.
  Interventions: Biological: R21 with Matrix-M1; Biological: ChAd63 ME-TRAP; Biological: MVA ME-TRAP
- Control Group 4a (No Intervention): These volunteers will not be vaccinated and will serve as infectivity controls when groups 1-3 undergo challenge.
- Control Group 4b (No Intervention): These volunteers will not be vaccinated and will serve as infectivity controls when group 5-7 and sterilely protected volunteers from groups 1-3 undergo challenge.
- Control Group 4c (No Intervention): These volunteers will not be vaccinated and will serve as infectivity controls if any volunteers from groups 5 and 7 are rechallenged.
- Fractional Dose (Group 5) (Active Comparator): R21 with Matrix-M1. Two vaccinations with 10 µg R21/ 50 µg Matrix-M1 on days 0 and 28 and one vaccination with 2µg R21/ 50 µg Matrix-M1 on day 56.
  Interventions: Biological: R21 with Matrix-M1
- Long-term Efficacy (Group 6) (No Intervention): Volunteers in this group have received vaccinations in a different malaria vaccine trial. These volunteers will not receive any vaccinations in this trial, but will undergo controlled human malaria infection as part of this study.
- Standard Dose x2 (Group 7) (Active Comparator): R21 with Matrix-M1. Two vaccinations with 10 µg R21/ 50 µg Matrix-M1 on days 0 and 28.
  Interventions: Biological: R21 with Matrix-M1

INTERVENTIONS:
Biological: R21 with Matrix-M1 — Vaccine
  Arms: Combination (Group 3); Fractional Dose (Group 5); High Dose (Group 2); Standard Dose x2 (Group 7); Standard Dose x3 (Group 1)
Biological: ChAd63 ME-TRAP — Vaccine
  Arms: Combination (Group 3)
Biological: MVA ME-TRAP — Vaccine
  Arms: Combination (Group 3)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of adjuvanted R21 alone and in combination with a viral-vectored vaccine regimen (constituting adjuvanted R21 + ChAd63 and MVA encoding ME-TRAP) against malaria sporozoite challenge in healthy malaria-naive volunteers.

Healthy adult volunteers will be recruited in London, Oxford and Southampton.

All vaccinations will be administered intramuscularly. The study involves having either two, three or five vaccinations and then undergoing challenge infection with malaria, or receiving no vaccinations then undergoing challenge infection with malaria.

DETAILED DESCRIPTION:
Vaccination phases and challenge procedures have been staggered over the trial period into 2 parts, challenges A and B.

Challenge A:

* Groups 1-3 consist of volunteers receiving either R21 alone or R21 + ChAd63-MVA ME-TRAP followed by CHMI by sporozoite challenge (mosquito bite) at week 12. Twelve volunteers will be recruited to each group.
* Group 4a will serve as infectivity controls, these volunteers will not be vaccinated.

Challenge B:

* Sterilely protected volunteers in groups 1 - 3 may be rechallenged to assess durability of efficacy, 5-12 months after the initial challenge.
* Groups 5-7 will also be enrolled to participate in challenge B.
* Group 5 (8 volunteers) will test the efficacy of standard dose R21 with a fractional third dose followed by CHMI at week 12.
* Group 6 will test the long-term efficacy of the standard dose R21 vaccination regimen (volunteers in this group will have already received their vaccinations whilst enrolled in the VAC053 malaria trial and will therefore not receive any additional vaccinations before undergoing challenge).
* Group 7 (8 volunteers) will test the efficacy of a two dose R21 vaccination regimen followed by CHMI at week 8.
* Group 4b will serve as infectivity controls for groups 5-7 and sterilely protected group 1-3 volunteers. Group 4c volunteers will be used as infectivity controls if any volunteers from groups 5 and 7 are rechallenged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception* for the duration of the study.
* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to take a curative anti-malaria regimen following CHMI.
* For volunteers not living close to their designated malaria challenge follow-up site (Oxford or Southampton): agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data as assessed by the investigator. If any volunteers in Group 1-3 undergo rechallenge, this exclusion criterion does not extend to the vaccines previously received in the VAC065 trial
* For Group 3 volunteers only: prior receipt of a non-malaria MVA or non-malaria adenovirus vectored experimental vaccine
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone
* Any clinical condition known to prolong the QT interval
* History of cardiac arrhythmia, including clinically relevant bradycardia
* Disturbances of electrolyte balance, eg, hypokalaemia or hypomagnesaemia
* Family history of congenital QT prolongation or sudden death
* Contraindications to the use of all three proposed anti-malarial medications; Riamet, Malarone and Chloroquine.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.60
* Positive family history in 1st and 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of adjuvanted R21 at two different doses and adjuvanted R21 + ChAd63 and MVA encoding ME-TRAP in healthy malaria-naïve volunteers as assessed by number of completely protected individuals. | 6 months
  Use statistical analysis to compare number of completely protected individuals (those who do not, by Day 21 following sporozoite challenge, develop blood stage infection measured by occurrence of P. falciparum parasitemia, assessed by blood slide) in the vaccine groups compared to the controls.
Safety of adjuvanted R21 at two different doses and adjuvanted R21 + ChAd63 and MVA encoding ME-TRAP in healthy malaria-naïve volunteers as assessed by frequency of adverse events. | 6 months
  Solicited and unsolicited adverse event data will be collected at each clinic visit from diary cards, clinical review, clinical examination (including observations) and laboratory results. This AE data will be tabulated and frequency, duration and severity of AEs compared between groups.

SECONDARY OUTCOMES:
Humoral immunogenicity generated in malaria naïve individuals with adjuvanted R21 at two different doses | 6 months
  Antibody response to the circumsporozoite protein generated by vaccination with adjuvanted R21.
Cell-mediated immunogenicity generated in malaria naïve individuals with ChAd63 and MVA encoding ME-TRAP | 6 months
  T-cell responses to the TRAP antigen of the malaria parasite generated by vaccination with ChAd63 and MVA encoding ME-TRAP .
Efficacy measured as time to P. falciparum parasitemia assessed by PCR against malaria sporozoite challenge, in healthy malaria-naïve volunteers. | 6 months
  Statistical analyses using blood stage infection as defined by 500 or more parasites/ml in peripheral blood by quantitative PCR.
Efficacy measured as time to P. falciparum parasitemia assessed by blood slide against malaria sporozoite challenge, in healthy malaria-naïve volunteers. | 6 months
  Statistical analyses using blood stage infection defined by a composite of symptoms, blood film result and parasitaemia.
Efficacy measured as time to P. falciparum parasitemia assessed by parasite density dynamics assessed by PCR against malaria sporozoite challenge, in healthy malaria-naïve volunteers. | 6 months
  Statistical analyses using blood stage malaria infection as defined by 20 or more P. falciparum parasites/ml in peripheral blood by quantitative PCR.

OTHER OUTCOMES:
Long term protective efficacy of adjuvanted R21 at two different doses and adjuvanted R21 + ChAd63 and MVA encoding ME-TRAP | 12 months
  Long term efficacy of the vaccination regimens will be assessed by re-challenging any sterilely protected individuals at 5 - 7 months after the first sporozoite challenge (~12 months after the start of the study) and comparing the number of re-challenges who develop blood stage infection with unvaccinated controls.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhil FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hosptal, Oxford, United Kingdom
Locations (3):
- United Kingdom (3):
  - NIHR Wellcome Trust Clinical Research Facility, Hammersmith Hospital, London
  - CCVTM, University of Oxford,, Oxford
  - Southampton National Institute for Health Research, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Venkatraman N, Silman D, Bellamy D, Stockdale L, Bowyer G, Edwards NJ, Griffiths O, Lopez FR, Powlson J, Mair C, Folegatti PM, Datoo MS, Morter R, Minassian AM, Poulton I, Collins KA, Brod F, Angell-Manning P, Berrie E, Brendish N, Glenn G, Fries L, Baum J, Blagborough AM, Roberts R, Lawrie AM, Angus B, Lewis DJM, Faust SN, Ewer KJ, Hill AVS. R21 in Matrix-M adjuvant in UK malaria-naive adult men and non-pregnant women aged 18-45 years: an open-label, partially blinded, phase 1-2a controlled human malaria infection study. Lancet Microbe. 2025 Mar;6(3):100867. doi: 10.1016/S2666-5247(24)00083-1. Epub 2025 Jan 10. PMID 39805301
- [Derived] Ssemaganda A, Giddam AK, Zaman M, Skwarczynski M, Toth I, Stanisic DI, Good MF. Induction of Plasmodium-Specific Immune Responses Using Liposome-Based Vaccines. Front Immunol. 2019 Feb 1;10:135. doi: 10.3389/fimmu.2019.00135. eCollection 2019. PMID 30774635